CLINICAL TRIAL: NCT03205085
Title: Determinants of Postoperative Right Heart Remodeling in Patients With Chronic Thrombo-Embolic Pulmonary Hypertension After Endarterectomy, or Pulmonary Arterial Hypertension After Lung Transplantation
Brief Title: Determinants of Right Heart Remodeling in Patients With CTEPH or PAH
Acronym: PRINCEPT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Chirurgical Marie Lannelongue (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2017-A00785-48
Record Dates: First submitted 2017-06-28; First posted 2017-07-02 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Chronic Thrombo-embolic Pulmonary Hypertension and Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Magnetic Resonance Spectroscopy; Blood Specimen Collection

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CTEPH PATIENTS (Experimental): Patients undergoing pulmonary endarterectomy for the treatment of chronic thromboembolic pulmonary hypertension (CTEPH).
  Interventions: Radiation: magnetic resonance imaging; Procedure: 2D and 3D trans-thoracic echocardiography; Other: Blood samples
- PAH PATIENTS (Experimental): patients with pulmonary arterial hypertension (PAH) undergoing lung transplantation
  Interventions: Radiation: magnetic resonance imaging; Procedure: 2D and 3D trans-thoracic echocardiography; Other: Blood samples

INTERVENTIONS:
Radiation: magnetic resonance imaging — assessment of right heart dimensions and function by cardiac magnetic resonance Imaging.
Procedure: 2D and 3D trans-thoracic echocardiography — assessment of right heart dimensions and function by 2D and 3D trans-thoracic echocardiography
Other: Blood samples — Blood samples for assays of immune inflammatory biomarkers (InterLeukin-18, CXCL9 or interferon

SUMMARY:
Right heart failure is the main cause of morbi-mortality in patients with pulmonary hypertension (PH), including patients of chronic thrombo-embolic pulmonary hypertension (CTEPH) or pulmonary arterial hypertension (PAH) etiologies. Endarterectomy is an effective treatment for patients with CTEPH to lower pulmonary pressure. Evidence of postoperative right heart remodeling are contrasted according to the studies and determinants of right heart failure are still unclear. Similarly, few evidence exists on right ventricular remodeling after bilateral lung transplantation for patients with pulmonary arterial hypertension (PAH). Recent evidence have supported the role of inflammation and immunity in the pathophysiology of PAH . While several cytokines have been shown to predict survival , little is known on the implication of inflammation and immunity in postoperative Right Ventricular failure in patients with PAH.

• The specific translational goal of this current project is to elucidate the role of immune biomarkers in 6 months postoperative right heart adverse remodeling in patients with CTEPH or PAH. We speculate that selected immune biomarkers (such as CXCL9, interleukin -18 or interferon) and growth factors (such as HGF) are correlated with mid-term postoperative right heart failure.

All consecutive adults with either CTEPH referred to our center for endarterectomy, or PAH referred for lung transplantation, will be included, aiming for 150 CTEPH and 50 PAH. After inclusion, patients will undergo assessment of right heart dimensions and function by cardiac magnetic resonance imaging (MRI, including 4-Dimensions blood flow sequences) and 2D and 3D trans-thoracic echocardiography (TTE), as well as immune panel analysis. All patients will undergo as part of routine care right heart catheterization within a week after TTE and MRI imaging. On the day of surgery, pulmonary pressure will be measured by right heart catheterization monitoring (as part of routine care) in order to estimate the drop of pressure and to adjust for the extent of endarterectomy for patients with CTEPH. TTE will also be performed on the day of surgery if possible. At 7 days post-endarterectomy or transplant, clinical outcomes will be collected and peripheral blood will be collected. Patients will be prospectively follow-up for 6 months. Death, need for reintervention, duration of vasopressor after surgery and number, duration and cause of readmission will be recorded. At 6 months after surgery, all survivors will undergo the same biological sampling, as well as an 4D MRI and a 2D and 3D TTE. Data of right heart catheterization at 6 months (as part of routine care) will be collected as well.

ELIGIBILITY:
Inclusion Criteria:

* adults (age > 18 years old)
* who give their informed consent for the protocol
* with either CTEPH referred to our insitution for pulmonary arterial endarterectomy. CTEPH is defined by invasive mean pulmonary arterial pressure ≥ 25mmHg at rest, secondary to chronic pulmonary embolism confirmed by computed tomographic (CT) angiography and/or ventilation/perfusion scan, according to the lastest guidelines
* Or with PAH referred to our institution for lung transplant. PAH is defined according to the latest guidelines by an invasive mean pulmonary arterial pressure ≥ 25mmHg, secondary to idiopathic, familial, drug or toxin, or connective tissue disease etiology.

Exclusion Criteria:

* pregnant women
* children
* congenital heart diseases
* contraindications for MRI such as metallic foreign bodies or devices, claustrophobia
* contraindication for surgery
* patients requiring preoperative mechanical assistance such as extracorporeal membrane oxygenation
* patients with pulmonary arterial sarcoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2017-08-09 (Actual); Primary Completion 2020-07-01 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
right ventricular adverse remodeling | 6 months
  postoperative right ventricular adverse remodeling, defined by increase above 10% in end-systolic right ventricular volume indexed on body surface area assessed by cardiac MRI.

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Marie Lannelongue, Le Plessis-Robinson, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dong ML, Azarine A, Haddad F, Amsallem M, Kim YW, Yang W, Fadel E, Aubrege L, Loecher M, Ennis D, Pavec JL, Vignon-Clementel I, Feinstein JA, Mercier O, Marsden AL. 4D flow cardiovascular magnetic resonance recovery profiles following pulmonary endarterectomy in chronic thromboembolic pulmonary hypertension. J Cardiovasc Magn Reson. 2022 Nov 14;24(1):59. doi: 10.1186/s12968-022-00893-x. PMID 36372884